CLINICAL TRIAL: NCT04074941
Title: The Effect of Sodium Reduction on Blood Pressure and Physical Function in Older Adults
Acronym: SOTRUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Shivani Sahni, Associate Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-2019-22
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Hypertension; Physical Disability; Aging
Keywords: Sodium Intake; Blood Pressure; Hypertension; Physical Function; Older Adults; Randomized Controlled Trial
MeSH Terms: conditions — Hypertension | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a low sodium diet or a usual sodium diet for a period of two weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study staff involved in administering the dietary intervention and assessing compliance will be masked to participants' outcome assessments (e.g. BP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low sodium diet (Experimental): This group will get a low sodium diet (<0.9 mg per kcal of energy intake).
  Interventions: Other: Dietary intervention
- Usual sodium diet (Active Comparator): This group will get a usual sodium diet (~2 mg per kcal of energy intake).
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Intervention include low sodium or usual sodium diet

SUMMARY:
This study will examine the effects of low sodium meal plan on seated blood pressure in older adults from a community-based, congregate senior living facility.

DETAILED DESCRIPTION:
Hypertension in older adults is a known contributor to both cardiovascular disease and falls. The Centers of Disease Control advocates for low sodium, senior meal plans as a strategy to lower blood pressure (BP). However, sodium is recommended to treat orthostatic hypotension (OH), a risk factor of falls. The long-term effects of low sodium intake on physical function are largely unknown in older adults.

The objective of this proposed pilot study is to determine the feasibility of an individual-level, randomized feeding study that examines the impact of sodium reduction on BP regulation among 40 semi-independent, older adults aged 60 and above.

Primary Aim 1: To determine the effects of a low sodium (<0.9 mg per kcal of energy intake), 2-week meal plan compared with a usual meal plan (average sodium ~2 mg per kcal of energy intake) on seated BP among independently living older adults.

Hypothesis Aim 1: Compared with the usual meal plan, a reduced sodium meal plan will lower seated BP in older adults after 2 weeks.

Feasibility Aim 1: To evaluate the recruitment experience, meal cost, meal delivery logistics, and compliance with and tolerability of the meal plan (urine sodium and palatability questionnaires).

Feasibility Aim 2: To determine effect size (variance) of secondary outcomes: standing BP, OH (standing minus seated BP), orthostatic symptoms, and a timed up and go test (TUG).

Eligible participants will be randomized to low versus usual sodium meal plans for two weeks. Assessments will be made at the in-person baseline visit, one week telephonic interview and 2 week in person follow-up visit.

The primary outcome is seated BP and secondary outcomes include orthostatic hypertension and Timed Up and Go (TUG) tests. Both primary and secondary outcomes will be measured twice: (1) before the study begins (baseline), and (2) after 2 week period. Patient-reported outcomes, dietary compliance, and urine electrolytes will be assessed as well.

Intent-to-treat analysis will be conducted for all endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Resident at Jack Satter House in Revere
* Age >= 60 years
* Resting systolic blood pressure 100-149 mm Hg and diastolic blood pressure <100 mm Hg
* Stable BP medications (no recent or intended changes)

Exclusion Criteria:

* Cognitive Impairment (Montreal Cognitive Assessment test <18)
* Unstable blood pressure medications in the past 2 months
* Terminal or mental illness
* Severe allergies to common foods
* Unwillingness to comply with the diet
* Physical inability to do a timed up and go test
* Active kidney dialysis or history of kidney transplant

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sahni, PhD, Principal Investigator — Marcus Institute, Hebrew SeniorLife and Harvard Medical School
Locations (1):
- Jack Satter House, Revere, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the approximately 285 residents of Jack Satter House, 59 adults expressed interest in participation. We ultimately enrolled 20 participants.
Period: Overall Study
Arm/Group | Low Sodium Diet | Usual Sodium Diet
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Sodium Diet | Usual Sodium Diet | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (6.1) | 79.6 (9.4) | 78.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Systolic blood pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 123.5 (9.7) | 121.1 (12.2) | 122.5 (10.7)
Diastolic blood pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 65.3 (11.1) | 62 (7.5) | 63.9 (9.5)
Hypertension, % [Count of Participants; unit: Participants] | 6 | 5 | 11
Hypertension medication use, % [Count of Participants; unit: Participants] | 7 | 5 | 12
Measured orthostatic hypertension, % [Count of Participants; unit: Participants] | 0 | 2 | 2
BMI, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (7.2) | 31.9 (7.9) | 32.1 (7.3)
Montreal Cognitive Assessment score [Mean (Standard Deviation); unit: scores on a scale] — Scores range from 0-30, with a score of 26 and higher generally considered normal
  scores on a scale | 24.3 (3.3) | 23.6 (1.9) | 23.9 (2.7)
Physical activity score [Mean (Standard Deviation); unit: scores on a scale] — Scores range from 0-42, with higher scores representing higher physical activity
  scores on a scale | 15.9 (15.1) | 22.8 (13.7) | 19.0 (14.5)
Timed-up-and-go, sec [Mean (Standard Deviation); unit: seconds] | 14.0 (6.2) | 13.4 (3.9) | 13.7 (5.1)
Estimated calorie intake, kcal/d [Mean (Standard Deviation); unit: kcal/day] | 1849 (244) | 1785 (311) | 1820 (270)

OUTCOME MEASURES:

1. Primary Outcome: Seated Blood Pressure
Description: Average of three seated systolic and diastolic blood pressure readings
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Sodium Diet | Usual Sodium Diet
Number analyzed (Participants) | 11 | 9
mmHg
  Follow-up seated systolic blood pressure | 112.1 (7.6) | 116.1 (13.0)
  Follow-up seated diastolic blood pressure | 60.3 (9.6) | 60.4 (8.0)

2. Secondary Outcome: Orthostatic Hypotension
Description: Measured from supine and standing systolic and diastolic blood pressure readings
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Sodium Diet | Usual Sodium Diet
Number analyzed (Participants) | 11 | 9
Participants | 3 | 5

3. Other Pre Specified Outcome: Timed up and go Test
Description: Participant will be asked to start from seated position, stand up from the chair, walk 3 meters in a straight line, turn, walk back to the chair and sit down. The investigators will use average of the two trials.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Low Sodium Diet | Usual Sodium Diet
Number analyzed (Participants) | 11 | 9
seconds | 13.8 (5.6) | 13.8 (4.9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Low Sodium Diet | Usual Sodium Diet
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Sodium Diet (N=11) | Usual Sodium Diet (N=9)
High blood glucose in participants with baseline diabetes (Endocrine disorders) | 0 (0) | 2 (2) — Self-reported

LIMITATIONS AND CAVEATS:
Limitations include low powered, which was expected as we fell short of recruitment goals and enrolled adults without elevated blood pressure. Our study lasted a short duration. Effects from sodium on BP may take up to 4 weeks, while effects on physical function may require even more time to occur. Our study included predominantly White obese females which limits generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT04074941/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT04074941/SAP_002.pdf
  • Informed Consent Form (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04074941/ICF_001.pdf